CLINICAL TRIAL: NCT05344014
Title: Evaluation of the Effect of the Photobiomodulation on the Efficacy of Anesthesia of Maxillary Permanent Molar Teeth With MIH
Brief Title: Anethesia Efficacy on Teeth With MIH (Molar Incisor Hypomineralisation)
Acronym: MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ulku Sermet Elbay, Assoc.Prof., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KAEK/04.bI.05
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Low-level-laser Theraphy; Anesthesia, Local; Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation group (Experimental): In the experimental group, before local infiltration anesthesia was administered, PBMT (a diode laser: 940 nm; continuous mode; 0.5W; 78 J/cm2) was applied perpendicular to the root surface at buccal and palatal area for 60 sec each).
  Interventions: Procedure: Photobiomodulation
- Placebo Group (Placebo Comparator): In the control group, the laser probe was directed to the mucosa for (buccal and palatal area), but not activated.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Photobiomodulation — In experimental groups, before topical anesthesia, PBMT was applied by utilizing a diode laser (EpiX; Biolase technology, inc., USA) with a continuous wavelength of 940 nm on a 400-μm fiber with only biostimulation properties. In accordance with the recommendations of the device's manufacturer, it was applied using circular motions in a manner as slowly as possible (an average of 33-36 circular movements in 60 s)
  Arms: Photobiomodulation group
Procedure: Placebo — In the control group (placebo), the laser probe was directed to the mucosa for (buccal and palatal area), but not activated, and the sound of the laser device previously recorded on the mobile telephone was played for the same time of experimental group in order to provide similar conditions
  Arms: Placebo Group

SUMMARY:
Difficulty in achieving anesthesia in teeth with molar incisor hypomineralisation (MIH) is a frequently reported clinical problem. The effect of low-level laser on the efficacy of anesthesia in teeth with MIH has not been studied yet. Aim of this study is to evaluate the effect of the Photobiomodulation on the efficacy of anesthesia of maxillary permanent molar teeth with MIH.

Design: The current study was conducted as a prospective, parallel-arm control, randomized, triple-blind clinical trial in children aged between 7to12 years. Maxillary permanent molar teeth with MIH requiring pulpotomy treatment were included. 70 participants were divided randomly into 2 groups as experiment (with PBMT) and control (Placebo) according to the anesthesia technique. In the experimental group, before local infiltration anesthesia was administered, PBMT (a diode laser: 940 nm; continuous mode; 0.5W; 78 J/cm2) was applied perpendicular to the root surface at buccal and palatal area for 60 sec each). In the control group, the laser probe was directed to the mucosa for (buccal and palatal area), but not activated. Evaluation of the pain scores were performed during the access cavity preparation of the pulpotomy treatment using the Face, Legs, Activity, Cry, Consolability (FLACC) Scale. Also, additional anesthesia requirements were assessed for both groups while working on the dentin and pulp

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Molar Incisor Hypoplasia (MIH)
* Maxillary permanent first molars with MIH
* Must be the score 3 of MIH (European Academy of Paediatric Dentistry MIH diagnostic criteria

Exclusion Criteria:

* The teeth showing irreversible pulp pathology (according to the American Association of Endodontics)
* The children who had negative or definitely negative behavior
* Allergy to local anesthetics
* Taking any medication that might affect the anesthetic assessment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluating efficacy of anesthesia with using the Face, Legs, Activity, Cry, Consolability (FLACC) Scale | Through study completion, an average of 24 weeks
  Anesthesia efficacy was evaluated objectively with the FLACC scale during the cavity preparation. Behavioral parameters were recorded during the cavity preparation (dentin cutting handpiece ) FLACC scale comprises of five sub-parameters. They are Face, Legs, Activity, Crying and Consolability. Each sub-parameter is given a pain score of 0 to 2. So total behavioral pain score range 0-10 as follows: 0 = relaxed and comfortable (no pain); 1-3= mild discomfort; 4-6 = moderate pain; and 7-10 = severe discomfort and/or pain. Success was achieved if patients experienced mild pain or no pain during the preparation of the cavity
Evaluating need of supplementary anesthesia | Through study completion, an average of 24 weeks
  The subjects with moderate/higher pain need supplementary anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Faculty of Dentistry, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Topcuoglu HS, Akpinar B. The effect of low-level laser therapy on the success rate of inferior alveolar nerve blocks in mandibular molars with symptomatic irreversible pulpitis: A randomized clinical trial. Int Endod J. 2021 Oct;54(10):1720-1726. doi: 10.1111/iej.13596. Epub 2021 Aug 2. PMID 34241896
- [Background] Ghabraei S, Chiniforush N, Bolhari B, Aminsobhani M, Khosarvi A. The Effect of Photobiomodulation on the Depth of Anesthesia During Endodontic Treatment of Teeth With Symptomatic Irreversible Pulpitis (Double Blind Randomized Clinical Trial). J Lasers Med Sci. 2018 Winter;9(1):11-14. doi: 10.15171/jlms.2018.03. Epub 2017 Dec 26. PMID 29399304
- [Background] Menoncin BLV, Portella PD, Ramos BLM, Assuncao LRDS, de Souza JF, Menezes JVNB. Dental anxiety in schoolchildren with molar incisor hypomineralization-A population-based cross-sectional study. Int J Paediatr Dent. 2019 Sep;29(5):615-623. doi: 10.1111/ipd.12503. Epub 2019 May 6. PMID 31009135